CLINICAL TRIAL: NCT01799577
Title: Comparison of 2-Dimensional and New Generation 3-Dimensional Laparoscopic Visions In An Experimental Model
Brief Title: Comparison of 2-Dimensional and 3-Dimensional Laparoscopic Visions
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BEHGynobs-4
Record Dates: First submitted 2013-02-13; First posted 2013-02-27 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Diagnostic Self Evaluation
Keywords: laparoscopy, accuracy, duration
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gynecologist: Gynecologist can use laparoscopic surgery.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — Two methods will be compare

SUMMARY:
This study tests the hypothesis that use of the 3-D laparoscopic vision system (Viking Systems, La Jolla, CA) can significantly improve technical ability on a complex laparoscopic tasks in an experimental model.

DETAILED DESCRIPTION:
7 tasks on a 3-D laparoscopic instrument fitted to the trainer box and subjective criteria (4 point lickert scale) were evaluated for this study. Totally twenty-four participants (8 experienced, 8 minimal experienced and 8 novices) were evaluated for different 10 tasks (touch the marked circle, pass the two circle with needle, pick-beads and place, grape the suture, move the needle from one instrument to another instrument, pick-and-place, cutting, three different suturing) in term of total task time and error number. Statistical Package Program was used to perform statistical analyses. The data were presented as arithmetic means and standard deviations were calculated in each group. A P value of <0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

medical doctors

Exclusion Criteria:

disabled person (about arms or vision problems)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Medical doctors
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
In order to test whether the 3-D laparoscopy vision system is superior or not than the 2-D laparoscopic vision system. | 15 days
  We want to test the 3-D laparoscopic vision system (Viking Systems, La Jolla, CA) can significantly improve technical ability on a complex laparoscopic tasks in an experimental model. 7 tasks on a 3-D laparoscopic instrument fitted to the trainer box and subjective criteria (4 point lickert scale) were evaluated for this study. Totally twenty-four participants (8 experienced, 8 minimal experienced and 8 novices) were evaluated for different 10 tasks in term of total task time and error number.

CONTACTS AND LOCATIONS:
Overall Officials: TANER USTA, M.D., Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Trainig and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Usta TA, Ozkaynak A, Kovalak E, Ergul E, Naki MM, Kaya E. An assessment of the new generation three-dimensional high definition laparoscopic vision system on surgical skills: a randomized prospective study. Surg Endosc. 2015 Aug;29(8):2305-13. doi: 10.1007/s00464-014-3949-0. Epub 2014 Nov 21. PMID 25414065